CLINICAL TRIAL: NCT00166010
Title: A Single-center, Pharmacokinetic Evaluation of Nesiritide in the Pediatric Population With Heart Failure
Brief Title: Effects of Nesiritide in Pediatric Patients With Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Observational study that DSMB placed on hold (withdrew 4 subjects). Protocol revised and received IND to become interventional PK study (no subjects enrolled).
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Janet Simsic, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003353
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure; Ventricular Dysfunction; Heart Decompensation
Keywords: drug; pediatrics; cardiac; Children with Cardiac Ventricular Failure
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nesiritide (Experimental)
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Standard dose of nesiritide which is a loading dose of 1 mcg/kg IV over 30 minutes followed by a nesiritide infusion at 0.01mcg/kg/min. All patients will be continually evaluated. At any time the attending physician may add or adjust treatment if deemed clinically indicated.

SUMMARY:
Children with severe heart failure need immediate appropriate care. New and better drugs are constantly being developed. As these drugs are approved for adult use, they are used off-label for children. The Food and Drug Administration (FDA) encourages clinical studies of drugs in children to further extend appropriate use of new medicines.

This study involves nesiritide, which was approved as a congestive heart failure treatment in adults in August 2001. The investigators' use of this drug in a pediatric population with severe heart failure has been encouraging. The investigators now wish to formally determine the pharmacokinetic and safety of Nesiritide in children.

The investigators will enroll 30 patients who are in the cardiac intensive care unit with severe heart failure. The data collected will include weights, vital signs, laboratory results, and echocardiography results. A research lab test called B-type natriuretic peptide (BNP) will be done several times during this study. If the patient still has an intravenous (IV) catheter, the blood sample will be taken from the IV. If the patient does not have an IV, the sample will be taken from a fingerstick.

The duration of the study will be the first 2 days of the patient's stay in the cardiac intensive care unit and thru discharge to evaluate the endpoint safety of Nesiritide. Additional information will also be collected if patient gets re-admitted within 30 days of discharge.

DETAILED DESCRIPTION:
Nesiritide (human recombinant B-type natriuretic peptide) has been recently approved by the Food and Drug Administration for the intravenous treatment of patients with decompensated congestive heart failure. Nesiritide has been studied in a broad range of patients, including the elderly, women, and African Americans, and patients with a history of various cardiovascular conditions including hypertension, diabetes, post myocardial infarction, atrial fibrillation/flutter, nonsustained ventricular tachycardia, left ventricular diastolic dysfunction, and acute coronary syndrome. However, clinical experience in the pediatric population has been limited.

Nesiritide is a human B-type natriuretic peptide (BNP) produced by recombinant technology having the same amino acid sequence as the naturally occurring human BNP. BNP is predominantly secreted by the cardiac ventricles in response to increased cardiac volume and pressure overload. Its pharmacologic effects include hemodynamic, neurohormonal, and renal. In adult studies, hemodynamic effects are characterized by balanced venous and arterial dilation, resulting in decreased preload and afterload demonstrated by a reduction of pulmonary capillary wedge pressure, pulmonary arterial pressure, and systemic vascular resistance while neurohormonal effects of nesiritide favorably inhibit the renin-angiotension-aldosterone system, leading to decreased plasma aldosterone and norepinephrine levels. The renal effects most often seen with nesiritide use is increased urine output and lower diuretic utilization.

There are currently no published articles discussing the use, including pharmacokinetics, of nesiritide in children. However, there are several centers that are currently using the drug - Columbus, Missouri; San Diego, California; Charleston, South Carolina; Loma Linda, California. Our experience in the infant after cardiac surgery and the older child with heart failure is encouraging. In children receiving nesiritide therapy, we noted significant clinical improvement with no appreciable side effects. Based on our initial experience, further prospective studies need to be performed in order to determine the pharmacokinetics and safety of using this therapy in the pediatric cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age newborn to 18 years.
2. Patients admitted to the CICU at Children's Healthcare of Atlanta in heart failure defined as decreased cardiac function and/or volume overload or admitted to the CICU at Children's Healthcare of Atlanta post-operatively after congenital heart defect repair surgery with increasing filling pressures and decreased ventricular compliance as seen by intracardiac line monitoring and echocardiography.
3. Receiving or about to receive nesiritide as medical therapy.
4. Informed consent will be signed by parent or guardian for all patients. (assent if applicable).

Exclusion Criteria:

1. Patients requiring extra corporeal membrane oxygenation (ECMO) support.
2. Patients requiring central veno-venous hemofiltration (CVVH).
3. Patients that are pregnant
4. Parent or legal guardian (or patient when applicable) refuses to sign informed consent.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine pharmacokinetics and safety of nesiritide in children | study period - first 2 days stay in cardiac intensive care unit thru hospital discharge and re-admission within 30 days of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Simsic, MD, Principal Investigator — Emory University

REFERENCES:
- [Background] Elkayam U, Akhter MW, Tummala P, Khan S, Singh H. Nesiritide: a new drug for the treatment of decompensated heart failure. J Cardiovasc Pharmacol Ther. 2002 Jul;7(3):181-94. doi: 10.1177/107424840200700308. PMID 12232567
- [Background] Marcus LS, Hart D, Packer M, Yushak M, Medina N, Danziger RS, Heitjan DF, Katz SD. Hemodynamic and renal excretory effects of human brain natriuretic peptide infusion in patients with congestive heart failure. A double-blind, placebo-controlled, randomized crossover trial. Circulation. 1996 Dec 15;94(12):3184-9. doi: 10.1161/01.cir.94.12.3184. PMID 8989127
- [Background] Abraham WT, Lowes BD, Ferguson DA, Odom J, Kim JK, Robertson AD, Bristow MR, Schrier RW. Systemic hemodynamic, neurohormonal, and renal effects of a steady-state infusion of human brain natriuretic peptide in patients with hemodynamically decompensated heart failure. J Card Fail. 1998 Mar;4(1):37-44. doi: 10.1016/s1071-9164(98)90506-1. PMID 9573502
- [Background] Mills RM, LeJemtel TH, Horton DP, Liang C, Lang R, Silver MA, Lui C, Chatterjee K. Sustained hemodynamic effects of an infusion of nesiritide (human b-type natriuretic peptide) in heart failure: a randomized, double-blind, placebo-controlled clinical trial. Natrecor Study Group. J Am Coll Cardiol. 1999 Jul;34(1):155-62. doi: 10.1016/s0735-1097(99)00184-9. PMID 10400005